CLINICAL TRIAL: NCT01391819
Title: An Epidemiological Study to Evaluate the Incidence, Clinical Characteristics and Economic Burden of Dengue in Brazilian Children
Brief Title: Study to Evaluate the Incidence, Clinical Characteristics and Economic Burden of Dengue in Brazilian Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 112994
Record Dates: First submitted 2011-07-08; First posted 2011-07-12 (Estimated); Results first posted 2017-04-26 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Dengue
Keywords: Brazil; Incidence; Dengue virus; Dengue; Dengue infection
MeSH Terms: conditions — Dengue | interventions — Data Collection

ARMS (1):
- Study cohort (Other): Children age 5 to 13 years at the time of enrollment, selected from schools in Fortaleza.
  Interventions: Other: Data collection; Procedure: Blood sample collection

INTERVENTIONS:
Other: Data collection — Socio-demographic information, medical history, yellow fever vaccination history and dengue suspicion data collection.
Procedure: Blood sample collection — A blood sample will be collected at each of the three scheduled study visits and any time during the study that dengue is suspected. Samples collected at scheduled visits will be tested for anti-dengue antibodies. Samples collected at visits for dengue suspicion will be tested for dengue diagnosis.

SUMMARY:
The aim of this study is to establish an active surveillance in order to generate dengue disease burden estimates including incidence rates, prevalence data, clinical presentation and cost of illness in Forteleza (Brazil).

DETAILED DESCRIPTION:
Prospective cohort study.

The study period initially planned to be two years, is extended by one year to cover one additional dengue season.

ELIGIBILITY:
Inclusion Criteria:

* Male or female between 5 and 13 years of age (including children at least 5 years of age and excluding children who reached their fourteenth birthday) at the time of enrollment.
* Written informed consent (and assent when applicable).
* Subjects who the investigator believes that they and/or their parent(s)/LAR can and will comply with the requirements of the protocol (e.g. willingness to do a hospital visit in case of dengue suspicion, willingness to attend the study hospital return for follow-up visits, able to observe for signs of dengue, understand how to take a temperature, etc).
* Subjects who plan to attend one of the study schools for two school years following enrollment.

Exclusion Criteria:

* Subjects planning to move from the study area during the two school years following enrollment.
* Child in care.
* Enrollment in another study that would conflict with the current study.

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2117 (Actual)
Dates: Start 2011-09-06 (Actual); Primary Completion 2015-01-30 (Actual); Study Completion 2015-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Fortaleza, Ceará, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] C B Coelho I, Haguinet F, B Colares JK, C B Coelho Z, M C Araujo F, Dias Schwarcz W, Duarte AC, Borges B, Minguet C, Guignard A. Dengue Infection in Children in Fortaleza, Brazil: A 3-Year School-Based Prospective Cohort Study. Am J Trop Med Hyg. 2020 Jul;103(1):100-111. doi: 10.4269/ajtmh.19-0521. Epub 2020 Apr 23. PMID 32342838

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 2117 subjects enrolled in the study, one subject was excluded due to protocol violation. Subjects attended 3 to 4 visits, during a 2 to 3 Year period: subjects enrolled in 2011-2012 who consented for participation of one additional year had 4 scheduled visits over 3 years, and those enrolled in 2013 had 3 scheduled visits over 2 years.
Groups:
- Dengue Group: Subjects, male and female, aged 5-13 years at the time of enrollment, enrolled for data collection and blood sampling for dengue evaluation, from Day 0 to Year 3.
Period: Overall Study
Arm/Group | Dengue Group
Started | 2116
Completed | 1714
Not Completed | 402
Not completed — Withdrawal by Subject | 56
Not completed — Migrated/moved from study area | 82
Not completed — Lost to Follow-up | 252
Not completed — Death | 3
Not completed — Other | 9

BASELINE CHARACTERISTICS:
Arm/Group | Dengue Group
Number analyzed (Participants) | 2116
Age, Continuous [Mean (Standard Deviation); unit: Years] | 8.997 (2.4637)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1096
  Male | 1020
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence of All Laboratory-confirmed Symptomatic Dengue Infection
Description: Laboratory-confirmed dengue infection refers to suspected symptomatic dengue cases with positive dengue virus identification or serologic evidence of dengue infection through dengue virus identification through Reverse Transcriptase quantitative Polymerase Chain Reaction (RT-qPCR) from first blood sample or anti-dengue Immunoglobulin type M/G (IgM/G) seroconversions between first and second blood sampling. Note: In the study report the denominator for incidence estimation has not been expressed as an absolute number of subjects, but in person-years. Therefore, the category "number of subjects analysed" has been populated with the number of enrolled subjects attended the study visit after the specified season and in each age stratum.
Time Frame: At Year 1 (2012)
Population: The analysis was performed on the According-To-Protocol (ATP) cohort, which included all subjects meeting all eligibility criteria of the study, with no elimination criteria during the study and complying with the procedures defined in the protocol.
Measure: Number (95% Confidence Interval); unit: Cases in 1000 person-years
Groups:
- Dengue 5-9Y Group: Subjects belonging to Dengue Group, male and female, aged 5-9 years at the time of the visit, enrolled for data collection and blood sampling for dengue evaluation.
- Dengue 10-17Y Group: Subjects belonging to Dengue Group, male and female, aged 10-17 years at the time of the visit, enrolled for data collection and blood sampling for dengue evaluation.
Arm/Group | Dengue 5-9Y Group | Dengue 10-17Y Group
Number analyzed (Participants) | 729 | 688
Cases in 1000 person-years | 10.5 [3.6 to 30.5] | 11.5 [0.1 to 1552.7]

2. Primary Outcome: Incidence of All Laboratory-confirmed Symptomatic Dengue Infection
Description: as for outcome 1
Time Frame: At Year 2 (2013)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Cases in 1000 person-years
Arm/Group | Dengue 5-9Y Group | Dengue 10-17Y Group
Number analyzed (Participants) | 818 | 932
Cases in 1000 person-years | 10.1 [2.3 to 44.9] | 25.8 [13.3 to 38.3]

3. Primary Outcome: Incidence of All Laboratory-confirmed Symptomatic Dengue Infection
Description: as for outcome 1
Time Frame: At Year 3 (2014)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Cases in 1000 person-years
Arm/Group | Dengue 5-9Y Group | Dengue 10-17Y Group
Number analyzed (Participants) | 576 | 1138
Cases in 1000 person-years | 3.9 [1.0 to 15.2] | 14.1 [-0.6 to 28.8]

4. Secondary Outcome: Proportion of Subjects With Prevalence of Past Dengue Infection (Dengue Seroprevalence) at Enrollment
Description: This outcome measures the occurrence of past dengue infections among subjects who had laboratory results. Proportion was estimated from logistic generalized estimating equations models (GEE) taking the clustering effect of the school into account and was presented per subject enrolment age. Immune response against dengue was assessed via Enzyme-linked Immunosorbent Assay (ELISA).
Time Frame: At Day 0 (At enrollment)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of subjects
Groups:
- Dengue Group: Subjects, male and female, aged 5-13 years at time of enrollment, enrolled for data collection and blood sampling for dengue evaluation, from Day 0 to Year 3.
Arm/Group | Dengue Group
Number analyzed (Participants) | 2104
Proportion of subjects
  IgG, 5 years old at enrollment: number analyzed (Participants) | 307
  IgG, 5 years old at enrollment | 32.57 [26.10 to 39.79]
  IgG, 6 years old at enrollment: number analyzed (Participants) | 240
  IgG, 6 years old at enrollment | 45.18 [42.86 to 47.51]
  IgG, 7 years old at enrollment: number analyzed (Participants) | 271
  IgG, 7 years old at enrollment | 38.86 [31.03 to 47.31]
  IgG, 8 years old at enrollment: number analyzed (Participants) | 267
  IgG, 8 years old at enrollment | 49.60 [37.39 to 61.85]
  IgG, 9 years old at enrollment: number analyzed (Participants) | 249
  IgG, 9 years old at enrollment | 50.20 [39.96 to 60.43]
  IgG, 10 years old at enrollment: number analyzed (Participants) | 247
  IgG, 10 years old at enrollment | 57.27 [49.42 to 64.78]
  IgG, 11 years old at enrollment: number analyzed (Participants) | 212
  IgG, 11 years old at enrollment | 68.87 [62.64 to 74.48]
  IgG, 12 years old at enrollment: number analyzed (Participants) | 185
  IgG, 12 years old at enrollment | 69.16 [61.56 to 75.84]
  IgG, 13 years old at enrollment: number analyzed (Participants) | 126
  IgG, 13 years old at enrollment | 70.16 [55.75 to 81.45]
  IgG, Total | 54.08 [46.59 to 61.40]

5. Secondary Outcome: Proportion of Subjects With Primary Asymptomatic Dengue Infection
Description: Asymptomatic dengue primary infection was defined as a documented seroconversion (anti-dengue IgG antibodies) between two sequential sera samples obtained during the scheduled visits, without suspicion of dengue. Proportion of asymptomatic dengue primary infection was analyzed among subjects who had no past dengue infection reported before the beginning of the period.
Time Frame: From Day 0 to Year 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: proportion of subjects
Arm/Group | Dengue Group
Number analyzed (Participants) | 1942
proportion of subjects
  Asymptomatic dengue, 2012: number analyzed (Participants) | 695
  Asymptomatic dengue, 2012 | 20.27 [13.63 to 29.07]
  Asymptomatic dengue, 2013: number analyzed (Participants) | 673
  Asymptomatic dengue, 2013 | 8.70 [6.88 to 10.94]
  Asymptomatic dengue, 2014: number analyzed (Participants) | 574
  Asymptomatic dengue, 2014 | 5.14 [4.40 to 6.01]
  Total | 13.09 [11.02 to 15.49]

6. Secondary Outcome: Number of Subjects With Laboratory Confirmed or Probable Dengue Cases According Symptomatic Dengue Definition (Primary, Secondary or Unknown) Among the Suspected Dengue Cases
Description: A case of primary or secondary symptomatic dengue infection was defined as laboratory confirmed or probable symptomatic dengue case whose previous sample collected at scheduled Visits 1- 4 (Day 0- Year 3) to detect anti-dengue IgG antibodies was seronegative or seropositive, respectively. A probable dengue case was defined as a suspected symptomatic dengue case with the following laboratory findings: -anti-dengue IgM or anti-dengue IgG positivity in at least one sample (in either blood sample 1 or 2) AND no evidence of viremia (negative dengue virus identification through RT-qPCR) in blood sample 1 AND no evidence of anti-dengue Ig M or IgG seroconversion between blood sample 1 and blood sample 2.
Time Frame: From Year 0 to Year 3
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Dengue Group
Number analyzed (Participants) | 188
Participants
  Primary, laboratory confirmed cases: number analyzed (Participants) | 42
  Primary, laboratory confirmed cases | 23
  Primary, probable cases: number analyzed (Participants) | 42
  Primary, probable cases | 19
  Secondary, laboratory confirmed cases: number analyzed (Participants) | 142
  Secondary, laboratory confirmed cases | 33
  Secondary, probable cases: number analyzed (Participants) | 142
  Secondary, probable cases | 109
  Unknown, laboratory confirmed cases: number analyzed (Participants) | 4
  Unknown, laboratory confirmed cases | 1
  Unknown, probable cases: number analyzed (Participants) | 4
  Unknown, probable cases | 3
  Total, laboratory confirmed cases | 57
  Total, probable cases | 131

7. Secondary Outcome: Incidence of All Laboratory-confirmed or Probable Symptomatic Dengue Infection
Description: Incidence of laboratory confirmed or probable symptomatic dengue infection was assessed by calendar year and age strata. Note: In the study report the denominator for incidence estimation has not been expressed as an absolute number of subjects, but in person-years. Therefore, the category "number of subjects analysed" has been populated with the number of enrolled subjects attended the study visit after the specified season and in each age stratum.
Time Frame: At Year 1 (2012)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Cases in 1000 person-years
Arm/Group | Dengue 5-9Y Group | Dengue 10-17Y Group
Number analyzed (Participants) | 818 | 1138
Cases in 1000 person-years | 30.3 [13.0 to 47.5] | 31.4 [14.8 to 48.1]

8. Secondary Outcome: Incidence of All Laboratory-confirmed or Probable Symptomatic Dengue Infection
Description: as for outcome 7
Time Frame: At Year 2 (2013)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Cases in 1000 person-years
Arm/Group | Dengue 5-9Y Group | Dengue 10-17Y Group
Number analyzed (Participants) | 818 | 1138
Cases in 1000 person-years | 56.7 [22.1 to 91.2] | 66.6 [40.0 to 93.2]

9. Secondary Outcome: Incidence of All Laboratory-confirmed or Probable Symptomatic Dengue Infection
Description: as for outcome 7
Time Frame: At Year 3 (2014)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Cases in 1000 person-years
Arm/Group | Dengue 5-9Y Group | Dengue 10-17Y Group
Number analyzed (Participants) | 818 | 1138
Cases in 1000 person-years | 13.6 [1.6 to 118.0] | 33.1 [10.0 to 56.2]

10. Secondary Outcome: Number of Dengue Infection Cases by Virus Type (DENV)
Description: Among virus types causing dengue infection were DENV-4 in 2012 and 2013 and DENV-1 in 2014, as assessed by PCR.
Time Frame: From Day 0 to Year 3
Population: as for outcome 1
Measure: Number; unit: Dengue infection cases
Arm/Group | Dengue Group
Number analyzed (Participants) | 21
Dengue infection cases
  DENV-4, 2012 | 8
  DENV-4, 2013 | 6
  DENV-1, 2014 | 7

11. Secondary Outcome: Number of Primary Laboratory Confirmed Symptomatic Dengue Infection Cases
Description: Primary symptomatic dengue infection cases are defined as laboratory confirmed symptomatic dengue cases whose previous sample collected at scheduled visits to detect anti-dengue IgG antibodies were seronegative. Analysis was done by calendar year and age strata. Note: In the study report the denominator for incidence estimation has not been expressed as an absolute number of subjects, but in person-years. Therefore the category "number of subjects analysed" has been populated with the number of enrolled subjects seronegative for anti-dengue IgG antibodies before the specified season and attended the study visit after the specified season, and in each age stratum.
Time Frame: At Year 1 (2012)
Population: as for outcome 1
Measure: Number; unit: Dengue infection cases
Arm/Group | Dengue 5-9Y Group | Dengue 10-17Y Group
Number analyzed (Participants) | 458 | 238
Dengue infection cases | 3 | 4

12. Secondary Outcome: Number of Primary Laboratory Confirmed Symptomatic Dengue Infection Cases
Description: as for outcome 11
Time Frame: At Year 2 (2013)
Population: as for outcome 1
Measure: Number; unit: Dengue infection cases
Arm/Group | Dengue 5-9Y Group | Dengue 10-17Y Group
Number analyzed (Participants) | 404 | 285
Dengue infection cases | 4 | 8

13. Secondary Outcome: Number of Primary Laboratory Confirmed Symptomatic Dengue Infection Cases
Description: as for outcome 11
Time Frame: At Year 3 (2014)
Population: as for outcome 1
Measure: Number; unit: Dengue infection cases
Arm/Group | Dengue 5-9Y Group | Dengue 10-17Y Group
Number analyzed (Participants) | 273 | 318
Dengue infection cases | 2 | 2

14. Secondary Outcome: Number of Secondary Laboratory Confirmed Symptomatic Dengue Infection Cases
Description: Secondary symptomatic dengue infection cases are defined as laboratory confirmed symptomatic dengue cases whose previous sample collected at scheduled visits to detect anti-dengue IgG antibodies were seropositive. Note: In the study report the denominator for incidence estimation has not been expressed as an absolute number of subjects, but in person-years. Therefore the category "number of subjects analysed" has been populated with the number of enrolled subjects seropositive for anti-dengue IgG antibodies before the specified season and attended the study visit after the specified season, and in each age stratum.
Time Frame: At Year 1 (2012)
Population: as for outcome 1
Measure: Number; unit: Dengue infection cases
Arm/Group | Dengue 5-9Y Group | Dengue 10-17Y Group
Number analyzed (Participants) | 268 | 450
Dengue infection cases | 4 | 3

15. Secondary Outcome: Number of Secondary Laboratory Confirmed Symptomatic Dengue Infection Cases
Description: as for outcome 14
Time Frame: At Year 2 (2013)
Population: as for outcome 1
Measure: Number; unit: Dengue infection cases
Arm/Group | Dengue 5-9Y Group | Dengue 10-17Y Group
Number analyzed (Participants) | 422 | 671
Dengue infection cases | 4 | 13

16. Secondary Outcome: Number of Secondary Laboratory Confirmed Symptomatic Dengue Infection Cases
Description: as for outcome 14
Time Frame: At Year 3 (2014)
Population: as for outcome 1
Measure: Number; unit: Dengue infection cases
Arm/Group | Dengue 5-9Y Group | Dengue 10-17Y Group
Number analyzed (Participants) | 300 | 824
Dengue infection cases | 0 | 10

17. Secondary Outcome: Number of Working Days Missed of Primary Care Giver 1 of Subjects With Laboratory Confirmed Symptomatic Dengue Cases
Description: The number of days off work from caregiver were recorded as part of health economics indirect resource utilization associated with symptomatic dengue infection.
Time Frame: From 21 up to 35 days post laboratory confirmed dengue onset
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Dengue Group
Number analyzed (Participants) | 12
Days | 2.4 (1.88)

18. Secondary Outcome: Number of Working Days Missed of Primary Care Giver 2 of Subjects With Laboratory Confirmed Symptomatic Dengue Cases
Description: as for outcome 17
Time Frame: From 21 up to 35 days post laboratory confirmed dengue onset
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Dengue Group
Number analyzed (Participants) | 4
Days | 1.8 (0.96)

19. Secondary Outcome: Number of Laboratory Confirmed Dengue Infection Cases Associated With Caregiver Absenteeism
Description: The number of laboratory confirmed dengue infections with primary caregivers missing from work was recorded as part of health economics indirect resource utilization associated with symptomatic dengue infection.
Time Frame: From 21 up to 35 days post laboratory confirmed dengue onset
Population: as for outcome 1
Measure: Number; unit: Dengue infection cases
Arm/Group | Dengue Group
Number analyzed (Participants) | 57
Dengue infection cases
  Primary care giver 1, Positive | 12
  Primary care giver 1, Negative | 42
  Primary care giver 1, Missing confirmed | 3
  Primary care giver 1, Not applicable | 0
  Primary care giver 2, Positive | 4
  Primary care giver 2, Negative | 46
  Primary care giver 2, Missing confirmed | 3
  Primary care giver 2, Not applicable | 4

20. Secondary Outcome: Number of School Days Missed by Subjects
Description: The number of school days missed by subjects due to dengue infection were recorded as part of the dengue active surveillance and indirect resource utilization associated with symptomatic dengue infection.
Time Frame: From 21 up to 35 days post laboratory confirmed dengue onset
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Dengue Group
Number analyzed (Participants) | 49
Days | 4.4 (2.58)

21. Secondary Outcome: Number of Laboratory Confirmed Dengue Infection Cases Associated With Subjects Absenteeism
Description: The number of laboratory confirmed dengue infection cases with subjects missing from school due to dengue infection were recorded as part of the dengue active surveillance and indirect resource utilization associated with symptomatic dengue infection.
Time Frame: From 21 up to 35 days post laboratory confirmed dengue onset
Population: as for outcome 1
Measure: Number; unit: Dengue infection cases
Arm/Group | Dengue Group
Number analyzed (Participants) | 57
Dengue infection cases
  Positive | 49
  Negative | 5
  Missing confirmed | 3
  Not applicable | 0

22. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: Serious adverse events (SAEs) were collected on the enrolled subjects. SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Day 0 to Year 3
Population: The analysis was performed on the Total cohort, which included all subjects enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Dengue Group
Number analyzed (Participants) | 2117
Participants | 0

23. Secondary Outcome: Number of Symptomatic Dengue Laboratory Confirmed Cases Associated With Hospitalization Direct Medical Resource
Description: Direct medical resource included hospitalization, stay in intensive care units (ICU), medications, diagnostic and therapeutic procedures
Time Frame: From Day 0 to Year 3
Population: as for outcome 1
Measure: Number; unit: Dengue infection cases
Arm/Group | Dengue Group
Number analyzed (Participants) | 57
Dengue infection cases
  Subject hospitalized, positive | 2
  Subject hospitalized, negative | 54
  Subject hospitalized, unknown | 1
  Hospitalized in a study hospital, positive | 1
  Hospitalized in a study hospital, negative | 1
  Hospitalized in a study hospital, unknown | 55

24. Secondary Outcome: Number of Hospitalization Days Due to Laboratory Confirmed Dengue Cases
Description: Length of hospitalization was part of the direct medical resource, associated with dengue infection.
Time Frame: From Day 0 to Year 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Dengue Group
Number analyzed (Participants) | 1
Days | 19.0 (0)

25. Secondary Outcome: Number of Dengue Infection Episodes - Clinical Symptom Since Onset of Suspected Dengue Cases: Temperature
Description: Temperature, expressed in degrees Celsius (°C), was among symptoms of symptomatic dengue infection.
Time Frame: From Day 0 to Year 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: °C
Arm/Group | Dengue Group
Number analyzed (Participants) | 55
°C | 37.18 (0.952)

26. Secondary Outcome: Number of Dengue Infection Episodes With Any Temperature Interval Since Onset of Suspected Dengue Cases, Among Laboratory Confirmed Dengue Cases
Description: Temperature intervals assessed varied from hypothermia 33.5 to 36.4 degrees Celsius (°C), to normal temperature 36.5-35.9 °C and hyperthermia 37 - 39.9 °C, or were unknown.
Time Frame: From Day 0 to Year 3
Population: as for outcome 1
Measure: Number; unit: dengue infection cases
Arm/Group | Dengue Group
Number analyzed (Participants) | 57
dengue infection cases
  33.5 - 33.9 °C | 0
  34 - 34.4 °C | 0
  34.5 - 34.9 °C | 0
  35 - 35.4 °C | 2
  35.5 - 35.9 °C | 2
  36 - 36.4 °C | 8
  36.5 - 36.9 °C | 11
  37 - 37.4 °C | 14
  37.5 - 37.9 °C | 7
  38 - 38.4 °C | 5
  38.5 - 38.9 °C | 4
  39 - 39.4 °C | 1
  39.5 - 39.9 °C | 1
  Unknown | 2

27. Secondary Outcome: Number of Laboratory Confirmed Dengue Episodes Associated With Clinical Symptoms
Description: Dengue related clinical symptoms included general symptoms, digestive symptoms, respiratory symptoms, hemorrhagic symptoms and any other signs among first symptoms.
Time Frame: From Day 0 to Year 3
Population: as for outcome 1
Measure: Number; unit: dengue infection cases
Arm/Group | Dengue Group
Number analyzed (Participants) | 57
dengue infection cases
  Headache | 43
  Retroorbital pain [eye pain] | 22
  Myalgia | 29
  Joint pain | 10
  Chills | 7
  Rash | 3
  Itching | 8
  At least one digestive sign among first symptoms | 38
  Abdominal pain | 17
  Nausea or vomiting | 29
  Diarrhea | 10
  At least one respiratory sign among first symptoms | 32
  Cough | 20
  Nasal congestion | 10
  Sore throat | 23
  Dyspnea | 0
  At least one hemorrhagic sign among first symptoms | 4
  Petechia | 3
  Purpura/ecchymosis | 0
  Hematemesis [vomiting of blood] | 1
  Melena/hematochezia [blood in stool] | 0
  Gingival bleeding | 0
  Epistaxis | 0
  Urinary tract bleeding | 0
  Unusual vaginal bleeding | 0
  At least one other signs among first symptoms | 33
  Pallor or cool skin | 2
  Conjunctivis | 2
  Lethargy or restlessness | 3
  Dizziness | 11
  Thoracic pain | 0
  Other | 28

ADVERSE EVENTS:
Time Frame: Serious Adverse Events were collected on the enrolled subjects throughout the study period (from Day 0 to Year 3).
Description: Adverse Events were not collected as blood sampling was the only invasive procedure performed.
Arm/Group | Dengue Group
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2117
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.